CLINICAL TRIAL: NCT01073423
Title: Improving Sleep and Quality of Life in Adults With HIV Disease: A Pilot Study
Brief Title: Improving Sleep and Quality of Life in Adults With HIV Disease
Acronym: R&R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kathryn A. Lee / Associate Dean of Research, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R&R Pilot
Record Dates: First submitted 2010-02-17; First posted 2010-02-23 (Estimated); Last update posted 2010-06-23 (Estimated); Status verified 2010-06

CONDITIONS: Insomnia
Keywords: HIV; sleep; insomnia; yoga; music
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Music Therapy; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental)
  Interventions: Behavioral: Yoga
- Music Therapy (Active Comparator)
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — 1-hour music therapy sessions, administered in group format 3 times per week for 8 weeks.
  Arms: Music Therapy
Behavioral: Yoga — 1-hour yoga sessions administered in group format 3 times per week for 8 weeks
  Arms: Yoga

SUMMARY:
The purpose of this study is to see if yoga or music therapy can improve the sleep of adults with HIV.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* HIV seropositive
* current sleep disturbance
* able to speak, read, and write in English
* a phone number to maintain contact with research team
* willing to provide copy of most recent CD4 and viral load values
* willing to wear actigraph for 1 week per month for 3 months
* willing to participate in group intervention sessions 3 times per week for 8 weeks

Exclusion Criteria:

* pregnancy
* psychiatric diagnosis, such as schizophrenia, dementia, bipolar disorder (depression not excluded)
* sleep disorder diagnosis, such as apnea or narcolepsy (insomnia not excluded)
* current yoga practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
self-reported sleep disturbance | 8 weeks

SECONDARY OUTCOMES:
actigraphic estimates of sleep quality and quantity | 8 weeks
self-reported well-being | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A. Lee, RN, PhD, Principal Investigator — University of California, San Francisco